CLINICAL TRIAL: NCT06019611
Title: A Pilot Study to Explore the Use of Percutaneous Spinal Stimulation in Participants With Multiple Sclerosis
Brief Title: Epidural Stimulation in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristin Zhao, PhD (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor-Investigator, Kristin Zhao, PhD, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-003967
Record Dates: First submitted 2023-08-02; First posted 2023-08-31 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis; Demyelinating Disorder; Autoimmune Diseases
MeSH Terms: conditions — Multiple Sclerosis; Demyelinating Diseases; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Percutaneous Epidural Stimulation (Experimental): Epidural spinal stimulation will be delivered via percutaneously implanted electrodes during rehabilitation. All implanted electrodes will be removed at the end of trial participation. The effects of epidural stimulation will be recorded via electrophysiological and biomechanical metrics described within the outcomes measures.
  Interventions: Device: Percutaneous epidural stimulation

INTERVENTIONS:
Device: Percutaneous epidural stimulation — Abbott percutaneous trial lead for epidural neurostimulation (Model 3086)
  Abbott clinician programmer for epidural and dorsal root ganglion neurostimulation (Model 3874)
  Ripple Neuromed Nomad Neurostimulation System

SUMMARY:
A study to quantify changes in motor performance of epidural stimulation in progressive multiple sclerosis (MS) patients over the course of 12 rehabilitation sessions.

DETAILED DESCRIPTION:
The purpose of this trial is to study spinal motor nerve response to electrical stimulation delivered directly to the epidural space, and to measure any changes in motor performance during 12 sessions over the course of one month.

ELIGIBILITY:
Inclusion Criteria:

* Myelopathy secondary to Progressive MS
* No clinical or radiologic MS relapses for > 5 years
* EDSS score of 6.5 (constant bilateral assistance required to walk about 20 meters without resting) as assessed by a Neurologist with a specialty in MS
* Able to ambulate 10 feet independently with or without gait aid use
* At least 22 years of age
* No changes to spasticity medications or dalfampridine over the last 3 months

Exclusion Criteria:

* Currently a prison inmate, or awaiting trial, related to criminal activity
* Pregnancy at the time of enrollment
* History of chronic and/or treatment resistant urinary tract infection
* Spasticity (grade of 4) measured bilaterally in two muscle groups using Modified Ashworth Scale (MAS). Muscle groups tested will include bilateral knee flexors, extensors; ankle plantarflexors, dorsiflexors
* Unhealed decubitus ulcer
* Unhealed skeletal fracture
* Receiving diathermy treatment
* Active participation in an interventional clinical trial
* Any illness or condition which, based on the research team's assessment, will compromise the patient's ability to comply with the protocol, patient safety, or the validity of the data collected during this study.
* History of coagulopathy or other significant cardiac or medical risk factors for surgery
* Ventilator-dependent respiration
* Diagnosed with cardiopulmonary dysfunction (e.g., chronic obstructive pulmonary disease, cardiac failure, or heart arrhythmia)
* Untreated clinical diagnosis of depression
* History of frequent hypotension characterized by light headedness, or loss of consciousness
* History of frequent hypertension characterized by headache, or bradycardia
* Any active, implanted medical device
* Treatment of chemodenervation and/or neurolysis during the trial, or within 6 months of initiating the trial

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 2 enrolled participants, 2 met inclusion criteria and proceeded to treatment.
Groups:
- Percutaneous Epidural Stimulation: Epidural spinal stimulation will be delivered via percutaneously implanted electrodes during rehabilitation. All implanted electrodes will be removed at the end of trial participation. The effects of epidural stimulation will be recorded via electrophysiological and biomechanical metrics described within the outcomes measures.
  Percutaneous epidural stimulation: Abbott percutaneous trial lead for epidural neurostimulation (Model 3086)
  Abbott clinician programmer for epidural and dorsal root ganglion neurostimulation (Model 3874)
  Ripple Neuromed Nomad Neurostimulation System
Period: Overall Study
Arm/Group | Percutaneous Epidural Stimulation
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Percutaneous Epidural Stimulation
Number analyzed (Participants) | 2
Age, Customized [Count of Participants; unit: Participants]
  Age 21 - 40 | 0
  Age 41+ | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Kinematics
Description: Change in maximum knee flexion, measured in degrees. Difference in maximum knee flexion between Baseline and End of Study with epidural stimulation off, and at End of Study between epidural stimulation off and epidural stimulation on.
Time Frame: Baseline and 4 weeks.
Measure: Mean (Full Range); unit: degrees
Arm/Group | Percutaneous Epidural Stimulation
Number analyzed (Participants) | 2
degrees
  Difference in maximum knee flexion between Baseline and End of Study with ES off | 15.5 [1 to 30]
  Difference in maximum knee flexion at End of Study between ES off and ES on | 10 [4 to 16]

2. Primary Outcome: Static Balance, Eyes-open.
Description: Percentage of change in postural sway area (cm^2) measured based on the center of force trajectory sway in the anterior-posterior and medial-lateral directions during static balance test with eyes-open. Decrease in postural sway area indicates an improvement in balance.
  Difference in postural sway area during balance test between Baseline and End of Study with epidural stimulation off, and at End of Study between epidural stimulation off and epidural stimulation on, both with subjects' eyes open, and closed.
Time Frame: Baseline and 4 weeks
Measure: Number; unit: percent change
Arm/Group | Percutaneous Epidural Stimulation
Number analyzed (Participants) | 2
percent change
  Difference in postural sway area between Baseline (ES off) and End of Study (ES off), eyes open | -50
  Difference in postural sway area between Baseline (ES off) and End of Study (ES off), eyes closed | -90
  Difference in postural sway area between End of Study (ES off) and End of Study (ES on), eyes open | -29
  Difference in postural sway area between End of Study (ES off) and End of Study (ES on), eyes closed | -54

3. Primary Outcome: Electromyography (EMG)
Description: Percentage of change in Root Mean Square (RMS) (time averaging, period of 0.25 sec) electromyography (EMG) (normalized to the max value during all gait cycles) of hamstring and rectus femoris during late-stance to mid-swing phase of gait, at End of Study between epidural stimulation on and epidural stimulation off.
Time Frame: End of Study (4 weeks)
Measure: Mean (Full Range); unit: percent change
Arm/Group | Percutaneous Epidural Stimulation
Number analyzed (Participants) | 2
percent change
  Change in voltage measurements of rectus femoris at End of Study, between ES on and ES off | -7 [-14 to 0]
  Change in voltage measurements of hamstring at End of Study, between ES on and ES off | 20 [0 to 40]

4. Primary Outcome: Spasticity, Knee Extensors (1)
Description: Change in measurements of the first swing angle (FSA) leg muscle tone utilizing Wartenberg's pendulum test, focusing on subject's most impaired side, measured at End of Study between epidural stimulation off and epidural stimulation on.
Time Frame: End of Study (4 weeks)
Measure: Mean (Full Range); unit: degrees
Arm/Group | Percutaneous Epidural Stimulation
Number analyzed (Participants) | 2
degrees | 6.5 [5 to 8]

5. Primary Outcome: Spasticity, Knee Extensors (2)
Description: Change in measurement of leg muscle tone utilizing the Modified Ashworth Scale (MAS). The Modified Ashworth Scale (MAS) is the standard clinical assessment tool for evaluating extremity spasticity in patients with central nervous system lesions. In this study, spasticity in the knee extensor muscles was assessed with the participant in a supine position, their legs dangling off the edge of an adjustable-height therapy mat. The resistance to knee flexion was graded on a 0-4 scale (0, 1, 1+, 2, 3, and 4) according to the MAS protocol for knee flexion, with lower scores indicating less muscle tone (0: no increase in muscle tone; 4: limb rigid in flexion).
  MAS was scored individually for both the right and left sides and reported separately at the end of the study, both with and without epidural stimulation. (A score of 1.5 indicates a MAS score of 1+).
Time Frame: End of Study (4 weeks)
Population: 1 participant analyzed per row.
Measure: Number; unit: score on a scale
Arm/Group | Percutaneous Epidural Stimulation
Number analyzed (Participants) | 2
score on a scale
  Participant 1, right side, ES off: number analyzed (Participants) | 1
  Participant 1, right side, ES off | 2
  Participant 1, right side, ES on: number analyzed (Participants) | 1
  Participant 1, right side, ES on | 1.5
  Participant 1, left side, ES off: number analyzed (Participants) | 1
  Participant 1, left side, ES off | 2
  Participant 1, left side, ES on: number analyzed (Participants) | 1
  Participant 1, left side, ES on | 0
  Participant 2, right side, ES off: number analyzed (Participants) | 1
  Participant 2, right side, ES off | 1.5
  Participant 2, right side, ES on: number analyzed (Participants) | 1
  Participant 2, right side, ES on | 1.5
  Participant 2, left side, ES off: number analyzed (Participants) | 1
  Participant 2, left side, ES off | 1.5
  Participant 2, left side, ES on: number analyzed (Participants) | 1
  Participant 2, left side, ES on | 1

6. Secondary Outcome: Overground Ambulation
Description: Change in walking speed during gait analysis, measured between Baseline and End of Study with epidural stimulation off, and at End of Study between epidural stimulation off and epidural stimulation on.
Time Frame: Baseline and 4 weeks
Measure: Mean (Full Range); unit: percent change
Arm/Group | Percutaneous Epidural Stimulation
Number analyzed (Participants) | 2
percent change
  Change in walking speed during gait analysis, measured between Baseline and End of Study with ES off | -25 [-32 to -18]
  Change in walking speed during gait analysis, measured at End of Study between ES off and ES on | 15 [6 to 25]

7. Secondary Outcome: Disability
Description: Measurement of changes in patient-reported disability status, utilizing the Short Form (36) Health Survey (SF-36). Questions are numerically ranked, with lower numbers representing more disability. Scores are combined into a composite scale from 0-100, with a score of zero equivalent to maximum disability and a score of 100 equivalent to no disability.
Time Frame: Baseline and 4 weeks
Population: 1 participant analyzed per row.
Measure: Number; unit: score on a scale
Arm/Group | Percutaneous Epidural Stimulation
Number analyzed (Participants) | 2
score on a scale
  Participant 1, Baseline: number analyzed (Participants) | 1
  Participant 1, Baseline | 68
  Participant 1, End of Study: number analyzed (Participants) | 1
  Participant 1, End of Study | 72
  Participant 2, Baseline: number analyzed (Participants) | 1
  Participant 2, Baseline | 56
  Participant 2, End of Study: number analyzed (Participants) | 1
  Participant 2, End of Study | 50

8. Secondary Outcome: Fatigue
Description: Measurement of changes in patient-reported fatigue status, utilizing the Modified Fatigue Impact Scale (MFIS). Items are scaled so that higher scores indicate a greater impact of fatigue on a person's activities. The total MFIS score can range from 0 to 84, with a score of zero equivalent to no fatigue and a score of 84 equivalent to maximum fatigue.
Time Frame: Baseline and 4 weeks
Population: 1 participant analyzed per row.
Measure: Number; unit: score on a scale
Arm/Group | Percutaneous Epidural Stimulation
Number analyzed (Participants) | 2
score on a scale
  Participant 1, Baseline: number analyzed (Participants) | 1
  Participant 1, Baseline | 30
  Participant 1, End of Study: number analyzed (Participants) | 1
  Participant 1, End of Study | 30
  Participant 2, Baseline: number analyzed (Participants) | 1
  Participant 2, Baseline | 30
  Participant 2, End of Study: number analyzed (Participants) | 1
  Participant 2, End of Study | 34

9. Secondary Outcome: Pain, Overall
Description: Measurement of changes in patient-reported pain status, utilizing the Pain Effects Scale (PES). Items are scaled so that higher scores indicate a greater impact of pain on a person's activities. The total PES score can range from 5 to 30, with a score of 5 equivalent to no pain and a score of 30 equivalent to maximum pain.
Time Frame: Baseline and 4 weeks
Population: 1 participant analyzed per row.
Measure: Number; unit: score on a scale
Arm/Group | Percutaneous Epidural Stimulation
Number analyzed (Participants) | 2
score on a scale
  Participant 1, Baseline: number analyzed (Participants) | 1
  Participant 1, Baseline | 17
  Participant 1, End of Study: number analyzed (Participants) | 1
  Participant 1, End of Study | 18
  Participant 2, Baseline: number analyzed (Participants) | 1
  Participant 2, Baseline | 19
  Participant 2, End of Study: number analyzed (Participants) | 1
  Participant 2, End of Study | 16

10. Secondary Outcome: Bladder Control
Description: Measurement of changes in patient-reported bladder control, utilizing the Bladder Control Scale (BLCS). Items are scaled so that lower scores indicate a greater degree of bladder control. The total BLCS score can range from 0 to 22, with a score of 0 equivalent to complete bladder control and a score of 22 equivalent to very poor bladder control.
Time Frame: Baseline and 4 weeks
Population: 1 participant analyzed per row.
Measure: Number; unit: score on a scale
Arm/Group | Percutaneous Epidural Stimulation
Number analyzed (Participants) | 2
score on a scale
  Participant 1, Baseline: number analyzed (Participants) | 1
  Participant 1, Baseline | 1
  Participant 1, End of Study: number analyzed (Participants) | 1
  Participant 1, End of Study | 0
  Participant 2, Baseline: number analyzed (Participants) | 1
  Participant 2, Baseline | 2
  Participant 2, End of Study: number analyzed (Participants) | 1
  Participant 2, End of Study | 13

11. Secondary Outcome: Bowel Control
Description: Measurement of changes in patient-reported bladder control, utilizing the Bowel Control Scale (BWCS). Items are scaled so that lower scores indicate a greater degree of bowel control. The total BWCS score can range from 0 to 26, with a score of 0 equivalent to complete bowel control and a score of 26 equivalent to very poor bowel control.
Time Frame: Baseline and 4 weeks
Population: 1 participant analyzed per row.
Measure: Number; unit: score on a scale
Arm/Group | Percutaneous Epidural Stimulation
Number analyzed (Participants) | 2
score on a scale
  Participant 1, Baseline: number analyzed (Participants) | 1
  Participant 1, Baseline | 1
  Participant 1, End of Study: number analyzed (Participants) | 1
  Participant 1, End of Study | 0
  Participant 2, Baseline: number analyzed (Participants) | 1
  Participant 2, Baseline | 5
  Participant 2, End of Study: number analyzed (Participants) | 1
  Participant 2, End of Study | 9

12. Secondary Outcome: Impact of Visual Impairment
Description: Measurement of changes in patient-reported visual impairment, utilizing the Impact of Visual Impairment Scale (IVIS). Items are scaled so that lower scores indicate less impairment on simple visual tasks. The total IVIS score can range from 0 to 15, with a score of 0 equivalent to no impairment and a score of 15 equivalent to severe visual impairment.
Time Frame: Baseline and 4 weeks
Population: 1 participant analyzed per row.
Measure: Number; unit: score on a scale
Arm/Group | Percutaneous Epidural Stimulation
Number analyzed (Participants) | 2
score on a scale
  Participant 1, Baseline: number analyzed (Participants) | 1
  Participant 1, Baseline | 3
  Participant 1, End of Study: number analyzed (Participants) | 1
  Participant 1, End of Study | 0
  Participant 2, Baseline: number analyzed (Participants) | 1
  Participant 2, Baseline | 0
  Participant 2, End of Study: number analyzed (Participants) | 1
  Participant 2, End of Study | 0

13. Secondary Outcome: Cognitive Dysfunction
Description: Measurement of changes in patient-reported cognitive dysfunction, utilizing the Perceived Deficits Questionnaire (PDQ). Items are scaled so that lower scores indicate less cognitive dysfunction. The total PDQ score can range from 0 to 80, with a score of 0 equivalent to no cognitive dysfunction and a score of 80 equivalent to extreme cognitive dysfunction.
Time Frame: Baseline and 4 weeks
Population: 1 participant analyzed per row.
Measure: Number; unit: score on a scale
Arm/Group | Percutaneous Epidural Stimulation
Number analyzed (Participants) | 2
score on a scale
  Participant 1, Baseline: number analyzed (Participants) | 1
  Participant 1, Baseline | 0
  Participant 1, End of Study: number analyzed (Participants) | 1
  Participant 1, End of Study | 0
  Participant 2, Baseline: number analyzed (Participants) | 1
  Participant 2, Baseline | 2
  Participant 2, End of Study: number analyzed (Participants) | 1
  Participant 2, End of Study | 9

14. Secondary Outcome: Mental Health
Description: Measurement of changes in patient-reported psychological distress and psychological well-being, utilizing the Mental Health Inventory (MHI-18). Items are scaled so that higher scores indicate less psychological distress. The raw score range is 0-100, with higher scores equivalent to less psychological distress and greater psychological well-being.
Time Frame: Baseline and 4 weeks
Population: 1 participant analyzed per row.
Measure: Number; unit: score on a scale
Arm/Group | Percutaneous Epidural Stimulation
Number analyzed (Participants) | 2
score on a scale
  Participant 1, Baseline: number analyzed (Participants) | 1
  Participant 1, Baseline | 78
  Participant 1, End of Study: number analyzed (Participants) | 1
  Participant 1, End of Study | 98
  Participant 2, Baseline: number analyzed (Participants) | 1
  Participant 2, Baseline | 73
  Participant 2, End of Study: number analyzed (Participants) | 1
  Participant 2, End of Study | 53

15. Secondary Outcome: Social Support
Description: Measurement of changes in patient-reported availability of social support, utilizing the Modified Social Support Survey (MSSS). Items are scaled so that higher scores indicate more social support. The total MSSS score can range from 18 to 90, with a score of 18 equivalent to no social support and a score of 90 equivalent to strong social support.
Time Frame: Baseline and 4 weeks
Population: 1 participant analyzed per row.
Measure: Number; unit: score on a scale
Arm/Group | Percutaneous Epidural Stimulation
Number analyzed (Participants) | 2
score on a scale
  Participant 1, Baseline: number analyzed (Participants) | 1
  Participant 1, Baseline | 66
  Participant 1, End of Study: number analyzed (Participants) | 1
  Participant 1, End of Study | 89
  Participant 2, Baseline: number analyzed (Participants) | 1
  Participant 2, Baseline | 63
  Participant 2, End of Study: number analyzed (Participants) | 1
  Participant 2, End of Study | 70

ADVERSE EVENTS:
Time Frame: 4 weeks.
Arm/Group | Percutaneous Epidural Stimulation
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Epidural Stimulation (N=2)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (2)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder incontinence (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT06019611/Prot_SAP_000.pdf